CLINICAL TRIAL: NCT05224830
Title: A Cross-sectional Study : Is There a Relationship Between Hyperventilation Syndrome and History of Acute SARS-CoV-2 Infection?
Brief Title: Relationship Between Hyperventilation Syndrome and SARS-CoV-2 Infection
Acronym: Hypercovid
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PI224-203
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Hyperventilation Syndrome
Keywords: covid-19; dyspnea; Hyperventilation Syndrome
MeSH Terms: conditions — COVID-19; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Presence of Hyperventilation Syndrome (HVS+): Study population was divided into two groups according to the diagnosis of Hyperventilation Syndrome HVS +- : Nijmegen questionnaire score > 23/64
  Interventions: Other: Nijmegen questionnaire score
- No presence of Hyperventilation Syndrome (HVS-).: Study population was divided into two groups according to the diagnosis of Hyperventilation Syndrome HVS - : Nijmegen questionnaire score < 24/64
  Interventions: Other: Nijmegen questionnaire score

INTERVENTIONS:
Other: Nijmegen questionnaire score — We collected the Nijmegen Questionnaire in order to diagnosis of Hyperventilation Syndrome

SUMMARY:
Following an acute COVID-19 infection, many patients suffer from long lasting physical symptoms that may greatly impair quality of life. Persisting dyspnea and other functional respiratory complaints could evoke Hyperventilation Syndrome (HVS) as a putative contributor of the long-COVID presentation in COVID-19 survivors. We aimed to assess the possible relationship between a HVS and previous acute SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Read and speak French
* Perform a pulmonary function test

Exclusion Criteria:

- incomplete questionnaire or inability to obtain an interpretable lung function assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion criteria were age greater than 18 years old, with the ability to perform a pulmonary function test in our Lung Function and Exercise Testing Department. Eligible patients were able to read and speak French in order to correctly answer to the self-reported questionnaire. The exclusion criteria were incomplete questionnaire or inability to obtain an interpretable lung function assessment.
Sampling Method: Non-Probability Sample
Enrollment: 2846 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Assess the relationship between a hyperventilation syndrome and previous acute SARS-CoV-2 infection. | Nijmegen questionnaire during 15 minutes (cross-sectional monocentric study)

SECONDARY OUTCOMES:
Assess the relationship between a hyperventilation syndrome and dyspnea | Nijmegen questionnaire during 15 minutes (cross-sectional monocentric study)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy., Vandœuvre-lès-Nancy, France